CLINICAL TRIAL: NCT02096848
Title: IDENTIFICATION OF THE EFFECT OF THE PNEUMOCOCCAL CONJUGATED VACCINE IN COSTA RICA
Brief Title: Microbiology of Otitis Media in Costarrican Children After PCV13 Introduction
Acronym: Microbiology
Status: Completed | Type: Observational
Sponsor: Instituto de Atención Pediátrica (Other)
Responsible Party: Principal Investigator, Arturo Abdelnour, MD Pediatric Inmunology, Instituto de Atención Pediátrica
Other Study IDs: Microbiology of Otitis Media
Record Dates: First submitted 2014-03-24; First posted 2014-03-26 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-09

CONDITIONS: Otitis Media in Children
Keywords: otitis media; microbiology; vaccines
MeSH Terms: conditions — Otitis Media

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bacteria isolated from children with otitis media
Oversight: Data Monitoring Committee: No

SUMMARY:
Studies which describe the bacterial aetiology and antimicrobial susceptibility in AOM children in Latin America are scarce. Interestingly, when the MEF microbiology was analyzed among 1,108 children aged 2-92 months with OM between years 2002 and 2007, non-typable H. influenzae was the most common pathogen isolated from the MEF of children with a otitis media failing to appropriate antimicrobial therapy.

PCV-7 (3 + 1 regimen) was introduced into the Costa Rican national immunization program in January 2009 and in August/September of 2011, it was changed for PCV 13 (-2+1 regimen). Following PCV-7 universal introduction in Costa Rica, between March of 2010 and January of 2011, MEF samples from Costa Rican children with OM, having received 0-4 PCV 7 vaccine doses, were obtained via tympanocentesis (88%) or from spontaneous otorrhoea (12%). It was interesting to observed that among the initial 134 OM episodes, the most common bacterial pathogen identified was H. influenzae (55%) followed by S. pneumoniae (31%) and that among the S. pneumoniae episodes, 55% were already non-PCV-7 serotypes and that 25% of these isolates were multi-drug resistant.

The primary objectives of the study are to analyze the effect of early universal utilization of PCV-13 in Costa Rican children with the number of H. influenzae and PCV-13- S. pneumoniae positive MEF cultures by comparing the data collected prospectively and by the same group of investigators that have collected the original data since 1992, from children for the post-PCV-13 introduction with anonymised information collected retrospectively pre-PCV-7 data (1999-2004) during a transition period in which PCV-7 was used in only the private settings (2005-2008) and during universal use of PCV-7 (2009-September 2011).

DETAILED DESCRIPTION:
Studies which describe the bacterial aetiology and antimicrobial susceptibility in AOM children in Latin America are scarce, however, since 1991, investigators in Costa Rica have follow the MEF microbiology of Costa Rican children with AOM including data before PCV 7, during a period of time when PCV-7 was used among high risk children and after universal introduction of a 3 + 1 PCV-7 regimen in Costa Rica. Published data from Costa Rican children with OM, collected between 1992 and 2007, describing the MEF microbiology indicated that overall S. pneumoniae was the most frequent pathogen followed by non-typable H. influenzae, M. catarrhalis and S. pyogenes. Interestingly, when the MEF microbiology was analyzed among 1,108 children aged 2-92 months with OM between years 2002 and 2007, non-typable H. influenzae was the mosto common pathogen isolated from the MEF of children with a otitis media failing to appropriate antimicrobial therapy.

PCV-7 (3 + 1 regimen) was introduced into the Costa Rican national immunization program in January 2009 and in August/September of 2011, it was changed for PCV 13 (-2+1 regimen). Following PCV-7 universal introduction in Costa Rica, between March of 2010 and January of 2011, MEF samples from Costa Rican children with OM, having received 0-4 PCV 7 vaccine doses, were obtained via tympanocentesis (88%) or from spontaneous otorrhoea (12%). It was interesting to observed that among the initial 134 OM episodes, the most common bacterial pathogen identified was H. influenzae (55%) followed by S. pneumoniae (31%) and that among the S. pneumoniae episodes, 55% were already non-PCV-7 serotypes and that 25% of these isolates were multi-drug resistant.

Based on the available information describing the worldwide modifications in the MEF microbiology of PCV-7 vaccinated children with OM (a proportional increase of cases caused by H. influenzae and non-PCV-7 S. pneumoniae serotypes), the primary objectives of the study are to analyze the effect of early universal utilization of PCV-13 in Costa Rican children with the number of H. influenzae and PCV-13- S. pneumoniae positive MEF cultures by comparing the data collected prospectively and by the same group of investigators that have collected the original data since 1992, from children for the post-PCV-13 introduction with anonymised information collected retrospectively pre-PCV-7 data (1999-2004) during a transition period in which PCV-7 was used in only the private settings (2005-2008) and during universal use of PCV-7 (2009-September 2011).

ELIGIBILITY:
Inclusion Criteria:

* All subjects must satisfy all the following criteria at study entry:

  * Age: more than 3 months and less than 6 years at the time of informed consent. The subject becomes ineligible at the seven birthday.
  * Signs and symptoms include:One of the functional or general signs of otalgia (or its equivalent: irritability), conjunctivitis, fever; AND EITHER Paradise's criteria (bulging, diffused or localised inflamed tympanic membranes) or Spontaneous otorrhoea of less than 24 hours.

Exclusion Criteria:

* Hospitalised during the diagnosis of otitis media or during treatment.
* Having an otitis externa, or otitis media with effusion
* Presence of a transtympanic tubes.
* Children presenting with a new episode of otitis media but having received antibiotic systemic therapy in the past 3 days for a separate illness.
* Receiving antimicrobial prophylaxis for recurrent acute otitis media.
* Received antibiotics for otitis media in the last day (exception: children with otitis media treatment failures must received antibiotic treatment within 3 to 5 days prior to study inclusion for the current otitis media episode).

Ages: 3 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged more than 3 months to less than 6 years, visiting with otitis media and from whom a middle ear fluid sample has been obtained.
  A cohort of children with the first episode of otitis media occurring before or at the age of 24 months of age and at least one month after completion of two doses of pneumococcal 13 valent vaccine will be followed until the participant completes 36 months of life.
Sampling Method: Non-Probability Sample
Enrollment: 387 (Actual)
Dates: Start 2012-05; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
• To compare the bacterial aetiology of middle ear fluid (MEF) samples collected from children with AOM following universal introduction of PCV-13 in the National Immunization Program of Costa Rica. | 3 years
  • To compare the bacterial aetiology of middle ear fluid (MEF) samples collected from children with AOM following universal introduction of PCV-13 in the National Immunization Program of Costa Rica.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Atencion Pediatrica, San José, Provincia de San José, Costa Rica

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arguedas A, Dagan R, Guevara S, Porat N, Soley C, Perez A, Brilla R. Middle ear fluid Streptococcus pneumoniae serotype distribution in Costa Rican children with otitis media. Pediatr Infect Dis J. 2005 Jul;24(7):631-4. doi: 10.1097/01.inf.0000168748.92510.45. PMID 15999006
- [Background] Abdelnour A, Soley C, Guevara S, Porat N, Dagan R, Arguedas A. Streptococcus pneumoniae serotype 3 among Costa Rican children with otitis media: clinical, epidemiological characteristics and antimicrobial resistance patterns. BMC Pediatr. 2009 Aug 14;9:52. doi: 10.1186/1471-2431-9-52. PMID 19682369